CLINICAL TRIAL: NCT04427462
Title: Linking Bioenergetic Phenotypes in Circulating Cells with Cardiometabolic Health in School-age Children
Brief Title: Bioenergetic Phenotypes and Cardiometabolic Health
Acronym: MI Energy
Status: Recruiting | Type: Observational
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 260376
Record Dates: First submitted 2020-04-10; First posted 2020-06-11 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2024-09

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood, urine, saliva, and stool will be collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This research study is about how daily activities, behaviors, and fitness affect the health and function of blood cells and their mitochondria, which are the powerhouses of the cells. These small mitochondria inside the cells make energy, and are very important for the health of the body.

DETAILED DESCRIPTION:
Determine the impact of physical activity and obesity status on circulating cells mitochondrial function (e.g., fat vs. carbohydrates combustion capacity, total oxidative capacity, mitochondrial number and proton leak).

ELIGIBILITY:
Inclusion Criteria:

Ages 8-10 years Boys and girls All ethnicity All BMI

Exclusion Criteria:

severe persistent asthma exercise induced asthma autism spectrum disorder attention deficit hyperactivity disorder attention deficit disorder

* Opposition defiant disorder
* conduct disorder
* epilepsy
* chronic kidney disease
* hormonal disease
* autoimmune diseases
* bleeding disorders
* chronic infections
* mental health disorder
* Type 2 and Type 1 diabetes
* Other pre-existing medical conditions or medications as determined by the investigators to affect the outcomes of interest

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 8-10 year olds
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Platelet mitochondrial respiration and its association with adiposity and peak aerobic capacity in children 8 to 10 years old. | 8 days
  Platelet mitochondrial respiration from isolated platelets will be measured using a flux analyzer. Adiposity will be measured with dual X-ray absorptiometry, and peak aerobic capacity with an incremental cycle ergometer test. measure physical activity

CONTACTS AND LOCATIONS:
Overall Officials: Elisabet Borsheim, Ph, Principal Investigator — Arkansas Children's Nutrition Center
Locations (1):
- Arkansas Children's Nutrition Center, Little Rock, Arkansas, United States